# A Gamified, Social Media Inspired Personalized Normative Feedback Alcohol Intervention for Sexual Minority Women

#### Consent Forms, Evaluation Study Invite, & Debriefing Statement

IRB approved on August 14<sup>th</sup>, 2018
Uploaded on May 5<sup>th</sup>, 2021

Trial Registration:ClinicalTrials.gov NCT03884478;

https://clinicaltrials.gov/ct2/show/NCT03884478

1. Competition Terms of Service & Privacy Policy (basic consent accepted prior to creating a user account in the LezParlay web app)

# TERMS OF SERVICE

#### **ELIGIBILITY**

To PARLAY you must identify as a lesbian, bisexual, or queer woman, be 21 years of age or older, and presently reside in the United States.

#### DATA USE, PRIVACY, & CONFIDENTIALITY

The LezParlay web application collects some personal data from its users. This information, detailed below, allows us assess interest from lesbian, bisexual, and queer women, understand app usage, and provide you with a smooth, efficient, and customized app experience. Personal data includes Facebook authentication data, demographic and other personally identifiable information that you voluntarily give to us when electing to create an account to participate in the LezParlay competition. When you register, you will sign-up with your email address and password or use your existing Facebook credentials. The only Facebook account data to be accessed by LezParlay is your email address and profile photo, and you will be prompted to grant or deny LezParlay permission to access these items. Next, you will create your LezParlay profile which includes your nickname/initials, age-group, sexual identity, and relationship status. Within the app, you will be represented by an optional photo and your public profile information (sexual identity, age-group, & relationship status will be visible to other authenticated players in the BROWSE area of the application, and the photos and public profiles of other users will similarly be visible to you in this area). However, you may choose to change your profile photo or delete it in the event you would prefer to remain faceless within the game by editing your account settings. You will also be prompted to provide a verifiable mobile phone number and email address when you create an account, however your contact information will remain private and will NOT be visible to other users. The app only uses this information to send you private results and prize notifications. You may opt out of receiving email and text notifications from LezParlay at any time, without penalty. To opt out of emails use the unsubscribe link provided. To opt out of text notifications simply reply too any text from LezParlay with "STOP". NONE of the information you provide at registration will be linked with your responses to competition questions or bets. Instead, your initial login at sign-up and the mobile phone number you provide will produce a unique code in our system which we will then use to link up your question responses, bets, and points across rounds. In sum, the application uses the personal data you provide to improve the user experience, facilitate representation and copresence among users, tailor your private results, and deliver these results to you. NONE of the personal data collected by the application will be shared with third parties under any circumstances. Derivative data includes information our servers automatically collect when you access the application, such as your actions that are integral to the application, including

responses to questions, points wagered, points scored, questions submitted, and question votes. Importantly, none of your actions in the app, including your answers to questions, or voting behavior will be view-able by other users accessing the application or shared with third parties. Data about the electronic device(s) and browsers you use to play LezParlay may also be logged by our server. This includes your device model, manufacturer, operating system, and browser version. This information is collected to improve the user experience on different devices and to aid us in troubleshooting should you report an issue using LezParlay on your device. Aggregated and de-identified personal, derivative, device/browser and analytics data may be analyzed by LezParlay project personnel in order to better understand application usage, determine the popularity of certain content, and inform future versions of the game. All data analysis and reporting for these purposes will focus on highlighting group trends rather than individual responses.

#### **DATA SECURITY**

LezParlay is an html5 web app that features the most advanced technologies and internal protocols (layered security, https protocol, SSL certificates, TSL encryption in transit, etc.) to transmit, secure, and store and protect application data. These protocols safeguard privacy between communicating applications and their users on the internet. Also used to secure bank and credit card transactions online, these protocols ensure that no third party may eavesdrop or tamper with submitted data.

#### POTENTIAL RISKS & BENEFITS

The risks associated with taking part in the competition lie in the potential for you to experience uncomfortable feelings due to the personal nature of some of the questions. Questions are somewhat edgy by design. They may ask, for example, how often you get drunk or have sex. You may choose to skip sensitive questions without penalty. However, we can only provide you points, scores, and detailed results corresponding to the questions you personally answer. You may also experience discomfort upon receipt of your detailed results. For example, it may be distressing to learn that other lesbians your age are drinking much less than you and exercising much more than you. You may opt out of receiving detailed feedback if you wish to do so. You may also choose to discontinue your participation in the competition at any time. This means if anything makes you feel too uncomfortable just quit playing! For some, participation in LezParlay may satisfy curiosities about LBQ communities or help to diminish harmful stereotypes. For others, learning about health and relationship behaviors of other lesbian and queer women may benefit their own health behaviors and relationships. Others may simply find entertainment in the wagers, scoring and results. De-identified, aggregated data collected by LezParlay may also help shape future programming by LezParlay community partners, which in turn, may benefit your future well-being.

#### **PRIZES**

The goal in LezParlay is to accumulate as many points as possible in each round and across rounds. You can earn points in each round by guessing and betting on the attitudes and behaviors of other LBQ women in your age-group and then reporting on your own attitudes & behaviors. In each round: a variable cash prize ranging from \$50 to \$500 will be awarded to the

player who scores the most points that round. In the event of ties, the top scorer who placed her bets earliest in the PARLAY period will be awarded the cash prize. After 7 rounds: Grand prizes will be awarded to the top 3 cumulative scorers in each age-group (20's, 30s, 40s, 50+) after all rounds have been played. In each age-group, first-place will receive \$1000, second place will receive \$500 and third place will receive \$250. In the event of ties, the cash prize will be awarded to the player who, on average across rounds played, placed her bets earliest.

## **GROUNDS FOR DISQUALIFICATION**

LezParlay is designed for lesbian, bisexual and queer-identified women living in the US of A. In effort to keep the game completely cis male and Russian bot free, users may be disqualified from the competition and have their account deleted if they appear to clearly NOT be an LBQ woman or residing in the US. Other grounds for disqualification include creating multiple accounts linked to different mobile numbers (in order to submit bets more than once each round) or attempting to cheat by any other means. In the spirit of healthy competition, we ask that you keep the detailed results you receive in the game private. This means not sharing any of the results you receive on social media or in private communication with friends until all rounds of the competition have been played. You may be disqualified if you violate this rule!

#### SUPPORT & TROUBLESHOOTING

If you experience trouble with the app on your mobile device or computer or are unable to login please email a description of your issue to support@lezparlay.com. Be sure to include the mobile phone number and email address associated with your LezParlay account so we can quickly fix any issues. We will shoot to resolve all issues within 24 hours.

#### ADDITIONAL INFORMATION

For additional information, questions about data usage, scoring, prizes, please contact Sarah Boyle, LezParlay's founder, at sarah@lezparlay.com or phone at 310.568.6681

2. Official Tester Invite Pop-Up Screen (End of Round 3 for eligible players)



3. Evaluation Study Informed Consent Form (End of Round 3 for eligible players interested in participating)



#### **PURPOSE**

LezParlay is grant-funded and we hope to apply for additional funds to continue the game in the future, add new features, improve the question topics and detailed results, and make future versions as enjoyable and beneficial as possible for lesbian, bisexual, and queer women. As such, the goals of this study are to: 1) evaluate the potential benefits associated with question topics and detailed results received in the LezParlay competition; and, 2) gather feedback on the player experience and areas in which the competition and app might be improved.

#### STUDY PARTICIPATION

Based on your verified status and participation in initial rounds of LezParlay, you have an opportunity to take part in this evaluation study as an Official Tester. Participation in the evaluation study involves playing remaining rounds of LezParlay and then completing a brief feedback survey about your experience in the competition following the final round of play. Each round of LezParlay will take no longer than 7 minutes to complete and the brief feedback survey will take no longer than 12 minutes to complete.

#### **INCENTIVES**

Official testers who complete remaining rounds of the competition (Completing Rounds 2 through 7) and submit the brief feedback survey at the end of the game will receive a \$60 in e-gift card of their choice (e.g., iTunes, Amazon, Target, Starbucks) to compensate them for their time and valuable insight. Importantly, as an Official Tester taking part in the evaluation study, you remain eligible for the cash prizes to be awarded to the competition's top scorers.

#### **DATA USE**

As a participant in the evaluation study, your demographic data, feedback survey data and responses to questions in LezParlay rounds may be aggregated with the responses of other

study participants and analyzed by the competition's founding psychologists at Loyola Marymount University. All research reports will de-identify all data from study participants and focus on highlighting group trends rather than individual responses.

#### CONFIDENTIALITY

While you may be visible and therefore potentially recognizable to other players in the game if you elect to upload a profile photo or bitmoji (as outlined in the app's Terms of Service and Privacy Policy), your participation in the Evaluation Study is completely confidential. There is no indication of which players are participating in the evaluation study and which are not. This means that no one will know you are participating in the evaluation study unless you tell them.

#### DATA SECURITY

As with all LezParlay data, feedback survey data is protected by Transport Layer Security (TLS) encryption (also known as HTTPS), which is a protocol that ensures privacy between communicating applications and their users on the internet. Also used to secure bank and credit card transactions online, TLS ensures that no third party may eavesdrop or tamper with submitted data.

#### POTENTIAL RISKS & BENEFITS

There are no additional risks associated with participation in the evaluation study beyond the personal nature of some of the questions to appear in LezParlay rounds and detailed results delivered in the game which may be distressing (As outlined in the Terms of Service and Privacy Policy you previously accepted). Benefits associated with evaluation study participation include the opportunity to share what you liked about LezParlay, what you disliked, and any ideas you may have about making it better with the competition's founders. In this way, you can help shape future versions of the competition and ensure that future versions are as satisfying and beneficial for you as possible.

Participation in the evaluation study is voluntary and you are free to stop participating at any time. To discontinue study participation, either simply stop playing LezParlay or email us at <a href="mailto:eval@lezparlay.com">eval@lezparlay.com</a> and let us know of your decision if you wish to no longer participate in the evaluation study but still wish to take part in the competition.

#### FOR MORE INFORMATION

If you have any questions or concerns about your participation in the evaluation study please contact the study's director, Sarah Boyle, on the campus of Loyola Marymount University, office phone number (310) 568-8661, email address sarah.boyle@lmu.edu If you have questions regarding your rights as a research participant, you may contact Dr. David Moffet, Chair of the Human Subjects Review Committee at Loyola Marymount

University, at (310) 338-4400 or <a href="mailto:david.moffet@lmu.edu">david.moffet@lmu.edu</a>. At the conclusion of this study, a summary of findings will be made publicly viewable at <a href="https://clinicaltrials.gov/ct2/show/NCT03884478">https://clinicaltrials.gov/ct2/show/NCT03884478</a>

### **PLEASE CHECK ONE OF THE BOXES BELOW:**

| By checking this box, I acknowledge that: • I have read and understood this informed consent information, and • I would like to participate in the LezParlay evaluation study |
|---|
| By checking this box, I acknowledge that: • I do not wish to participate in the LezParlay evaluation study. |

# 4. Debriefing Statement (presented following the post competition feedback survey)



Thanks again for helping us evaluate LezParlay! Before you go we wanted to give you some more information about the detailed results you received in the LezParlay as an Official Tester. In addition to getting your feedback and ideas for the next version of the competition, another goal of this study was to evaluate whether delivering results for health-related topics in LezParlay had any benefits for players' health and well-being. To fully examine this, we had to make sure that balanced groups of Official Testers received more and less health-related feedback.

So, full disclosure, the topics you received detailed results on in Rounds 3 and 4 of the game were not totally random in the same way they were in all of the other rounds (where they were determined by the doors you chose to open). Instead, as an Official Tester you were randomized to receive a specific sequence of feedback in Rounds 3 and 4 and the doors you selected were fixed to open to either health-related topics or topics unrelated to health. So, we're not sure if the health-related detailed results were beneficial yet, but analyzing the data from this study will allow us to find out! We also plan to examine whether you all reported different types of psychological benefits and/or differential levels liking for aspects of the competition based on the sequences of detailed results you received.

If you are interested in finding out what we learn here please let us know by sending an email to sarah@lezparlay.com and we'll be sure to send you a summary of results when they are ready. Thanks again for your participation!